CLINICAL TRIAL: NCT07249944
Title: Myofunctional Therapy for Children With Obstructive Sleep Apnoea - a Multi-centre Randomised Controlled Trial
Brief Title: Myofunctional Therapy for Children With OSA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other); Kwong Wah Hospital (Other); United Christian Hospital (Other); Queen Mary Hospital, Hong Kong (Other); The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kate Ching Ching Chan, Associate Professor, Department of Paediatrics, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MFTOSA
Record Dates: First submitted 2025-10-01; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: Children; Obstructive sleep apnoea; Myofunctional therapy; Randomised controlled trial; Intervention
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Myofunctional Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomisation procedures will be performed by research personnel blinded to the participants' characteristics and independent of the data collection and analysis. While it is not possible to blind the participants to their group assignment, the outcome assessor, who is independent of randomisation and study procedures, will be blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will undergo a MFT programme with telemedicine support.
  Interventions: Behavioral: Myofunctional therapy
- Controls (No Intervention): Participants in the control group will receive standard care, such as anti-inflammatory medications if indicated, without the Myofunctional therapy .

INTERVENTIONS:
Behavioral: Myofunctional therapy — Myofunctional therapy (MFT) has been proposed as an adjunctive therapy for obstructive sleep apnoea (OSA) in children. Some studies have reported improved sleep parameters and reduced oral breathing after MFT.
  Arms: Intervention group

SUMMARY:
Myofunctional therapy (MFT) has been proposed as an adjunctive therapy for obstructive sleep apnoea (OSA) in children.

Some studies have reported improved sleep parameters and reduced oral breathing after MFT. However, the level of evidence in these studies is limited, with most being case series or case-control studies. There have been only a few randomised controlled trials (RCTs), and these studies have had limitations such as low response rate, short follow-up periods, and the existing evidence does not adequately address the potential clinical benefits and the impact on craniofacial structure. Additionally, there is a lack of evidence regarding the effectiveness of additional measures, such as remote guidance and supervision, in improving treatment outcomes in children. Therefore, there is a need for further research to address these gaps and provide more robust evidence on the efficacy of MFT in children with OSA. The objective of this study is to investigate the efficacy of MFT in children with OSA through a multi-centre randomised controlled trial (RCT). 174 children aged 6-12 years old with OSA will be recruited and randomly assigned to either the intervention or control group. All children will undergo standardised evaluation at baseline and follow-up visits. In the intervention arm, a 24-week myofunctional therapy targeting orofacial MFT, breathing, and postural re-education, with incorporation of telemedicine for remote training and monitoring. In the control arm, children will receive standard care without MFT. The primary outcome measure will be obstructive apnoea hypopnoea index measured by polysomnography. Secondary outcome measures will be the oral breathing pattern, OSA-related symptoms, and quality of life. The treatment effect on outcomes will be examined using a mixed-effects model with an intention-to-treat approach. Subgroup analyses will explore potential effect modification by important participant characteristics, such as OSA severity and compliance. This study will generate evidence-based information regarding the efficacy of MFT in children with OSA and will inform clinical practice.

DETAILED DESCRIPTION:
Myofunctional therapy (MFT) has been proposed as an adjunctive therapy for obstructive sleep apnoea (OSA) in children. Some studies have reported improved sleep parameters and reduced oral breathing after MFT. However, the level of evidence in these studies is limited, with most being case series or case-control studies. There have been only a few randomised controlled trials (RCTs), and these studies have had limitations such as low response rate, short follow-up periods, and absence of polysomnographic measurement after intervention. Moreover, the existing evidence does not adequately address the potential clinical benefits and the impact on craniofacial structure. Additionally, there is a lack of evidence regarding the effectiveness of additional measures, such as remote guidance and supervision, in improving treatment outcomes in children. Therefore, there is a need for further research to address these gaps and provide more robust evidence on the efficacy of MFT in children with OSA.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6-12 years, with this age range, children start to have a greater ability to understand and follow instructions, making them more likely to comply and cooperate with the treatment procedures, and at the same time this age range remains a critical and modifiable developmental window when interventions can address underlying orofacial muscle and respiratory muscle dysfunctions and enhance the potential for long-term benefits.
2. Diagnosed with OSA based on clinical evaluation and polysomnography (oAHI ≥ 1/hour). The clinical evaluation will involve assessing the presence of habitual snoring, which is defined as snoring occurring 3 nights or more per week on average as reported by parents or caregivers, and any of the following features suggestive of SDB such as oral breathing, respiratory pauses, observed apnoeas, or increased work of breathing during sleep. Children with persistent OSA, documented by repeat PSG, can be included after receiving standard treatments (such as adenotonsillectomy treatment).
3. Informed consent from a parent or a legal guardian.

Exclusion Criteria:

* Genetic, syndromal, or metabolic disease
* Congenital or acquired neuromuscular disease
* Syndromal craniofacial abnormalities or previous craniofacial surgery
* Severe developmental delay (developmental or functional age <66% of chronological age)
* Children with OSA who are indicated for and will receive other treatments such as adenotonsillectomy, positive airway pressure therapy or orthodontic treatment.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 174 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
oAHI measured by PSG | 24 weeks
  oAHI measured by PSG

SECONDARY OUTCOMES:
Presence of oral breathing | 24 weeks
  Presence of oral breathing
Symptoms of sleep-disordered breathing | 24 weeks
  Pediatric Sleep Questionnaire
Daytime sleepiness | 24 weeks
  Modified Epworth Sleepiness Scale
OSA specific quality of life | 24 weeks
  OSA-18 questionnaire
Child behavioural and emotional measures | 24 weeks
  Child Behaviour Checklist
Lip and tongue strength and endurance | 24 weeks
  Lip and tongue strength and endurance measured using the Iowa Oral Performance Instrument
Free tongue length | 24 weeks
  Free tongue length measured using the Quick Tongue-tie Assessment Tool from the insertion of the lingual frenulum to the tongue tip
Tongue mobility | 24 weeks
  Tongue mobility measured by Mpal/Mmax, where Mpal and Mmax refer to the maximal distance between incisors when the tongue tip touches the palatal papilla and during whole mouth opening, respectively
Photogrammetry | 24 weeks
  Craniofacial landmarks will be located and recorded as pixel coordinates on the image following established procedures. Measurements of craniofacial linear distances, angles, and upper body posture will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ching Ching, Kate CHAN, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided